CLINICAL TRIAL: NCT06216015
Title: Exercise Training in Kidney Transplant Recipients (EXTRA Trial) Evaluating Physiological and Molecular Outcomes
Brief Title: Exercise Training and Kidney Transplantation
Acronym: EXTRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo de Luca Correa (Other)
Collaborators: Catholic University of Brasília (Other); Federal University of São Paulo (Other)
Responsible Party: Sponsor-Investigator, Hugo de Luca Correa, Principal Investigator, Catholic University of Brasília
Organization: Catholic University of Brasília (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 50129315.2.0000.5505
Record Dates: First submitted 2024-01-01; First posted 2024-01-22 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Solid Organ Transplant Rejection; Chronic Kidney Failure; Quality of Life; Inflammation; Muscle Weakness
Keywords: Exercise training; Nephrology; Transplantation; Chronic kidney disease; Exercise physiology; Quality of life
MeSH Terms: conditions — Kidney Failure, Chronic; Inflammation; Muscle Weakness; Renal Insufficiency, Chronic | interventions — Exercise; Exercise Therapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Exercise training group (Experimental): The training programs will encompass three phases, with a gradual progression in both intensity and duration. Each phase will span a duration of four weeks, culminating in a comprehensive 24-week training regimen.
  Interventions: Other: Exercise training
- Control group (No Intervention): Control group will continue their usual care without exercise interventions.
- Continue exercise (Active Comparator): Following the 24-week training regimen, patients will have the option to decide whether they wish to continue their exercise training. This group will include individuals who choose to persist with their exercise routine.
  Interventions: Other: Continue exercising
- Discontinue exercise (Active Comparator): Following the 24-week training regimen, patients will have the option to decide whether they wish to continue their exercise training. This group will comprise individuals who opted not to continue their exercise routine.
  Interventions: Other: Discontinue exercising

INTERVENTIONS:
Other: Exercise training — Participants will engage in combined training five times a week, with activities including 2 minutes of stationary marching and a set of 15 repetitions for squats, bilateral hip abduction, plantar flexion, floor abdominal exercises, and arm flexion with the knee close to the ground. Additionally, twice a week on non-consecutive days, volunteers partake in 20 minutes of aerobic walking.
  The second program starts with a 2-minute stationary march, followed by 2 sets of 12 repetitions for free squats, hip abduction, plantar flexion, stiff-legged deadlifts, arm flexion with knee support, floor abdominal exercises, and concludes with 30 minutes of aerobic exercise.
  The third program starts with a 2-minute stationary march, followed by 3 sets of 12 repetitions for free squats, hip abduction, plantar flexion, stiff-legged deadlifts, arm flexion, floor abdominal exercises, and includes thrice-weekly aerobic sessions lasting 30 minutes each.
  Other Names: Exercise therapy; Exercise; Combined exercise
  Arms: Exercise training group
Other: Continue exercising — Following the 24-week training regimen, patients will have the option to decide whether they wish to continue their exercise training. This group will include individuals who choose to persist with their exercise routine.
  Arms: Continue exercise
Other: Discontinue exercising — Following the 24-week training regimen, patients will have the option to decide whether they wish to continue their exercise training. This group will comprise individuals who opted not to continue their exercise routine.
  Arms: Discontinue exercise

SUMMARY:
The goal of this clinical trial is to investigate the physiological and molecular effects of exercise training in transplant recipients. The main questions it aims to answer are:

1. Can exercise training improve physical fitness and muscle strength in transplant recipients?
2. Can exercise training modulate inflammatory profile, hormones, lipid profile, and exercise-induced molecules in transplant recipients?
3. Can exercise training improve blood pressure and endothelial health in transplant patients?

Participants will be invited to an exercise training program 6-month after their transplant surgery. Body composition, physical assessment, and blood draw will be assessed at baseline and 24-weeks after exercise or control regimen.

Researchers will compare exercise group vs. routine care group to see if exercise training impact the health-related outcomes of this population.

DETAILED DESCRIPTION:
The study will involve inviting participants to join an exercise training program six months after their transplant surgery. The research will include baseline assessments and measurements, such as body composition, physical assessment, and blood draws. These assessments will be conducted both at the beginning of the study and 24 weeks after participants have undergone either the exercise regimen or a control regimen.

The research team will compare two groups: the exercise group and the routine care group. The goal is to examine whether participating in an exercise training program has a significant impact on various health-related outcomes in transplant recipients when compared to individuals receiving standard care.

This clinical trial seeks to understand the potential benefits of exercise training on physical fitness, quality of life, inflammatory and molecular profiles, as well as cardiovascular health in individuals who have undergone organ transplantation. The comparison between the exercise group and the routine care group will provide valuable insights into the effectiveness of exercise interventions for this specific population.

ELIGIBILITY:
Inclusion Criteria:

* Medical Authorization:
* Stable Health Status
* Medication Consistency
* No History of Severe Cardiovascular Events
* No Major Orthopedic Issues
* Non-Smokers or Consistent Smoking Habits
* Ability to Comply with Study Protocols

Exclusion Criteria:

* Inability to Comply
* Cognitive disorders
* Unwillingness to Continue
* Unstable Health Conditions
* Physical limitations during the protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 345 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Functional performance | Baseline, after 24-weeks and at the end of the protocol
  6-minute walking test
Muscle strength | Baseline, after 24-weeks and at the end of the protocol
  One Repetition Maximum Test
Isometric muscle strength | Baseline, after 24-weeks and at the end of the protocol
  Handgrip strength
Physical fitness | Baseline, after 24-weeks and at the end of the protocol
  Ergospirometric Test

SECONDARY OUTCOMES:
Inflammatory profile | Baseline, after 24-weeks and at the end of the protocol
  Interleukin 6, interleukin 10, and tumor necrosis factor
Urea-to-creatinine ratio | Baseline, after 24-weeks and at the end of the protocol
  Urea and creatinine will be combined to report urea-to-creatinine ratio
Blood glucose | Baseline, after 24-weeks and at the end of the protocol
  Fasting blood glucose levels
Hormones | Baseline, after 24-weeks and at the end of the protocol
  Irisin, Klotho, and adiponectin
Graft rejection | Through study completion, an average of 2 years
  Number of patients that rejected their graft

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in exercise and transplantation. Data or samples shared will be coded. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).